CLINICAL TRIAL: NCT05039112
Title: Clinical Comparison of 2 Daily Disposable Toric Soft Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: CLA306-E001
Record Dates: First submitted 2021-08-31; First posted 2021-09-09 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: Refractive Errors; Astigmatism
Keywords: Contact lenses; Daily disposable
MeSH Terms: conditions — Refractive Errors; Astigmatism

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- P1fA, then MyDay Toric (Other): Verofilcon A toric contact lenses worn first, with stenfilcon A toric contact lenses worn second, as randomized. Each product will be worn bilaterally (in both eyes) for 8 (-0/+3) days in a daily disposable modality.
  Interventions: Device: Verofilcon A toric contact lenses; Device: Stenfilcon A toric contact lenses
- MyDay Toric, then P1fA (Other): Stenfilcon A toric contact lenses worn first, with verofilcon A toric contact lenses worn second, as randomized. Each product will be worn bilaterally (in both eyes) for 8 (-0/+3) days in a daily disposable modality.
  Interventions: Device: Verofilcon A toric contact lenses; Device: Stenfilcon A toric contact lenses

INTERVENTIONS:
Device: Verofilcon A toric contact lenses — Soft contact lenses for optical correction of astigmatism, used as indicated
  Other Names: PRECISION1 for Astigmatism; P1fA
Device: Stenfilcon A toric contact lenses — Soft contact lenses for optical correction of astigmatism, used as indicated
  Other Names: MyDay Toric

SUMMARY:
The purpose of this study to evaluate the overall performance of PRECISION1™ for Astigmatism contact lenses with MyDay® Toric contact lenses.

DETAILED DESCRIPTION:
Subjects will be expected to attend 4 visits and wear study lenses daily for approximately 10 hours per day. On the day prior to the Week 1 Follow-up visit of each crossover period, subjects will be asked to wear the respective study lens for at least 16 hours. The expected duration of subject participation in the study is approximately 3 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

* Successful wear of toric soft contact lenses in both eyes for a minimum of 5 days per week and 10 hours per day during the past 3 months.
* Willing to wear study contact lenses for at least 16 hours on the day prior to the Week 1 Follow up visit of each lens type.
* Other protocol-defined inclusion criteria may apply.

Key Exclusion Criteria:

* Current/previous wear of PRECISION1 for Astigmatism or MyDay Toric contact lenses.
* Current wear of spherical contact lenses.
* Wears habitual contact lenses in an extended wear modality (routinely sleeping in lenses for at least 1 night per week).
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2021-11-29 (Actual)

PRIMARY OUTCOMES:
Percent of lenses with axis orientation within ±30 degrees inclusive from the intended axis, 10 minutes after lens insertion | Day 1, 10 minutes after lens insertion, each product
  Axis orientation (orientation of the scribe mark) will be assessed by slit lamp examination and recorded as deviations from intended axis.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, Vision Care, Study Director — Alcon Research, LLC
Locations (6):
- United States (6):
  - Alcon Investigator 6565, Maitland, Florida
  - Alcon Investigator 6567, Pittsburg, Kansas
  - Alcon Investigator 8097, Sterling Heights, Michigan
  - Alcon Investigator 6313, Powell, Ohio
  - Alcon Investigator 6401, Warwick, Rhode Island
  - Alcon Investigator 6353, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No